CLINICAL TRIAL: NCT01784874
Title: Immunogenicity of the Purified Vero Rabies Vaccine - Serum Free in Comparison With the Human Diploid Cell Vaccine, Imovax® Rabies in Pre-exposure Use in Healthy Adults
Brief Title: Comparison of Purified Vero Rabies Vaccine, Serum Free With Human Diploid Cell Vaccine in Pre-exposure Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VRV02; U1111-1124-7459 (Other: WHO)
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Rabies
Keywords: Rabies; Human Diploid Cell Vaccine; Imovax® Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purified Vero Rabies Vaccine Group (Experimental): Participants will receive the Purified Vero Rabies Vaccine (VRVg) Serum Free
  Interventions: Biological: Purified Vero Rabies Vaccine (VRVg) - Serum Free
- Imovax® Rabies Vaccine Group (Experimental): Participants will receive the Imovax® Rabies
  Interventions: Biological: Imovax® Rabies: inactivated rabies vaccine

INTERVENTIONS:
Biological: Purified Vero Rabies Vaccine (VRVg) - Serum Free — 0.5 mL, Intramuscular
  Arms: Purified Vero Rabies Vaccine Group
Biological: Imovax® Rabies: inactivated rabies vaccine — 1.0 mL, Intramuscular
  Other Names: Imovax® Rabies
  Arms: Imovax® Rabies Vaccine Group

SUMMARY:
The aim of this study is to generate data on immunogenicity and safety of Purified Vero Rabies Vaccine - Serum Free (VRVg) in comparison with Imovax® Rabies in order to support the registration of VRVg in the USA.

Primary Objectives:

* To demonstrate that VRVg is non inferior to Imovax® Rabies in terms of proportion of subjects achieving an rabies virus neutralizing antibody (RVNA) titer ≥ 0.5 IU/mL at Day 42.
* To demonstrate that the observed proportion of subjects achieving an RVNA titer ≥ 0.5 IU/mL at Day 42 is at least 99%, with a 95% lower confidence limit of at least 97%.

Secondary Objectives:

* To assess the clinical safety of VRVg each vaccine after each vaccine injection when administered in a pre-exposure schedule.
* To describe the immune response induced by each vaccine 21 days after two vaccinations (Day 28) in a randomized subset of subjects and 14 days after the last vaccination of the primary vaccination series.
* To describe antibody persistence at 6 and 12 months after the first vaccination in all subjects, and at 18 and 24 months in a subset of subjects.

DETAILED DESCRIPTION:
The vaccination will be given in three injections, at Day 0, Day 7, and Day 28, respectively, based on the Advisory Committee on Immunization Practice (ACIP) and the World Health Organization (WHO) recommendations for pre-exposure regimen. A booster dose will be administered 1 year after the first vaccine injection in a randomized subset of participants.

Safety will be assessed in all participants up to 28 days after vaccination, as applicable, in terms of occurrence of adverse events (AEs), and serious adverse events (SAEs) and adverse events of special interest (AESIs) up to Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to < 65 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and comply with all trial procedures.

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after last vaccination)
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination)or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks following any trial vaccination
* Previous vaccination against rabies (in pre- or post-exposure regimen) with either the trial vaccine or another vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
* At high risk for rabies exposure during the trial
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a vaccine containing any of the same substances as the vaccines used in the study
* Self-reported thrombocytopenia, contraindicating intra muscular (IM) vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4°F). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* History of Guillain-Barré Syndrome.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 408 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with rabies virus neutralizing antibody (RVNA) titer ≥ 0.5 IU/mL at Day 42 (14 days after the last vaccination of primary vaccination series). | Day 42 post-vaccination
  Rabies virus neutralizing antibody titer will be determined by the rapid fluorescent focus inhibition test (RFFIT)
Antibody Persistence in terms of rabies virus neutralizing antibody titers at 6 months and 12 months after the first vaccination | 6 and 12 months post-vaccination
  Rabies virus neutralizing antibody titer will be determined by the rapid fluorescent focus inhibition test (RFFIT)

SECONDARY OUTCOMES:
Number of Participants Reporting Solicited Injection Site Reactions, Solicited Systemic Reactions, Unsolicited Systemic Reactions, and Serious Adverse Events Occurring Throughout the Trial | Day 0 up to 12 months post-vaccination
  Solicited injection site reactions: pain, erythema, and swelling. Solicited systemic reactions: fever (temperature), headache, malaise, and myalgia.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (6):
- United States (6):
  - Redding, California
  - Sacramento, California
  - Omaha, Nebraska
  - Austin, Texas
  - Fort Worth, Texas
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Pichon S, Moureau A, Petit C, Chu L, Essink B, Muse D, Saleh J, Guinet-Morlot F, Minutello AM. Safety and immunogenicity of a serum-free purified Vero rabies vaccine in healthy adults: A randomised phase II pre-exposure prophylaxis study. Vaccine. 2022 Aug 5;40(33):4780-4787. doi: 10.1016/j.vaccine.2022.06.040. Epub 2022 Jun 28. PMID 35778281
- See also: Related Info — http://www.sanofipasteur.com